CLINICAL TRIAL: NCT05316233
Title: Multicenter, Evaluator-blinded, Randomized, Controlled Study of the Safety and Effectiveness of JUVÉDERM® VOLITE™ XC Injectable Gel for Improvement in Neck Appearance
Brief Title: A Study to Assess Adverse Events and Change in Disease Activity of JUVÉDERM® VOLITE™ XC Injectable Gel for Change in Neck Appearance in Adult Participants
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2029-701-008
Record Dates: First submitted 2022-03-31; First posted 2022-04-07 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: Neck Lines

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- VOLITE XC (Experimental): Participants will receive VOLITE XC for initial treatment and followed for up to 14 Months. Participants will have the opportunity to receive optional touch-up and optional repeat treatment of VOLITE XC during the follow-up duration period.
  Interventions: Device: VOLITE XC
- Control Group (Other): The control group received no treatment and will be followed for up to 6 months after randomization. Participants can then opt to receive VOLITE XC and followed for 6 Months.
  Interventions: Device: VOLITE XC

INTERVENTIONS:
Device: VOLITE XC — Intradermal Injection
  Other Names: JUVÉDERM® VOLITE™ XC
Device: VOLITE XC — Subdermal Injection
  Other Names: JUVÉDERM® VOLITE™ XC

SUMMARY:
The cumulative effect of aging and environmental exposures (ie, ultraviolet, infrared, and visible light radiation and pollution) leads to wrinkles, discoloration, laxity, and roughness of sun exposed skin. The neck is a frequently mentioned area by patients complaining about its crepey texture and deep lines. VOLITE XC is a crosslinked HA gel implant formulated with lidocaine that was developed to provide a safe, minimally invasive method of treating fine lines and improving skin quality. The purpose of this study is to assess adverse events and effectiveness of VOLITE XC in adults seeking improvement in neck appearance.

VOLITE XC is an investigational product being developed for the improvement of horizontal neck lines. Participants are placed in 1 of 2 groups, called treatment arms. There is a 1 in 3 chance that participants will be assigned to the control group. Around 212 adult participants with transverse neck lines will be enrolled in the study at approximately 20 sites.

Participants in the treatment group will receive VOLITE XC at Day 1 and followed for up to 14 Months. Participants will have the opportunity to receive optional touch-up and optional repeat treatment of VOLITE XC during the follow-up duration period. The control group received no treatment and will be followed for up to 6 months after randomization. Participants can then opt to receive VOLITE XC and followed for 6 Months.

There may be higher treatment burden for participants in this trial compared to their standard of care. Participants will attend regular visits during the study at a hospital or clinic. The effect of the treatment will be checked by medical assessments, checking for side effects and completing questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Participants in general good health as determined by Treating Investigator's judgment, including no known active pandemic infection.
* Participants seeking improvement of transverse neck lines.
* Has moderate or severe transverse neck lines (ATNLS Grade 2 or 3) on EI live assessment.

Exclusion Criteria:

* Neck deformity or significant skin laxity with severe redundant folds.
* Significant skin pigmentation disorders or discoloration in the neck area that would interfere with the visual assessment of the neck area.
* Current cutaneous inflammatory or infectious processes (eg. acne, herpes), abscess, an unhealed wound, or a cancerous or precancerous lesion on the neck.
* Tendency to develop hypertrophic scarring.
* History of thyroid cancer, skin cancer of the neck, radiation of the treatment area, or de novo cancer in the treatment area.
* Permanent soft tissue fillers in the neck area.
* Semi-permanent soft tissue fillers in the neck area within 2 years before enrollment.
* HA fillers or autologous fat in the neck area within 12 months before enrollment.
* Mesotherapy, photomodulation, intense pulsed light, radiofrequency, dermabrasion, chemical peel, microneedling, laser, or other cosmetic procedures in the neck area within 12 months before enrollment.
* Botulinum toxin in the neck area within 6 months before enrollment.
* Deoxycholic acid injections or cryolipolysis in the submentum area within 6 months before enrollment.
* Neck surgeries and procedures.
* Neck tattoos, piercings, pigmentation, hair, or past trauma that would interfere with the visualization of the neck area for the effectiveness assessments.
* Pregnant, nursing or planning a pregnancy.

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 159 (Actual)
Dates: Start 2022-05-02 (Actual); Primary Completion 2024-09-12 (Actual); Study Completion 2024-09-12 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants Achieving "Responder" status based on Evaluating Investigator's (EI) live assessment of transverse neck lines using the Allergan Transverse Neck Lines Scale (ATNLS) | Month 1
  A "responder" is a participant with at least 1-grade improvement on the ATNLS. ATNLS is a 5-point photonumeric scale to grade the severity of transverse neck lines (0=None, 4=Extreme)
Number of Participants with Adverse Events | Up to 14 Months
  An adverse event (AE) is defined as any untoward medical occurrence in a participant or clinical investigation participant administered a pharmaceutical product which does not necessarily have a causal relationship with the treatment. The investigator assesses the relationship of each event to the use of study drug.

SECONDARY OUTCOMES:
Percentage of Participants Achieving "Responder" Status for EI's Assessment of global aesthetic improvement on the neck using the Global Aesthetic Improvement Scale (GAIS) | Month 1
  A "responder" is a participant who shows improvement in the overall aesthetic assessment on the neck using GAIS. GAIS is a 5-point ordinal scale (2=Much Improved, -2=Much Worse).
Percentage of Participants Achieving "Responder" Status for Participant's Assessment of global aesthetic improvement on the Neck using GAIS | Month 1
  A "responder" is a participant who shows improvement in the overall aesthetic assessment in the neck using GAIS. GAIS is a 5-point ordinal scale (2=Much Improved, -2=Much Worse).
Change from baseline to Month 1 in the Rasch-transformed scores on FACE-Q Appraisal of the Neck questionnaire | Baseline to Month 1
  FACE-Q is a 10-item questionnaire assessing various aspects of the neck appearance. In the FACE-Q Appraisal of the Neck questionnaire, the responses will be summed and converted to a Rasch-transformed score that ranges from 0 to 100.

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (15):
- United States (15):
  - Steve Yoelin MD Medical Associate Inc /ID# 239072, Newport Beach, California
  - Laser & Skin surgery Medical group, Inc /ID# 241999, Sacramento, California
  - Cosmetic Laser Dermatology /ID# 239121, San Diego, California
  - Art of Skin MD /ID# 239071, Solana Beach, California
  - Center for Dermatology and Dermatologic Surgery /ID# 239137, Washington D.C., District of Columbia
  - Hevia Cosmetic Dermatology /ID# 239118, Coral Gables, Florida
  - Skin Research Institute LLC /ID# 239109, Coral Gables, Florida
  - Research Institute of the Southeast, LLC /ID# 239070, West Palm Beach, Florida
  - Delricht Research /ID# 242001, New Orleans, Louisiana
  - Rkmd, Llc /Id# 239075, North Bethesda, Maryland
  - image Dermatology, P.C. /ID# 239136, Montclair, New Jersey
  - Skin And Aesthetics Surgery Of Manhattan /ID# 243607, New York, New York
  - Mariwalla Dermatology /ID# 239102, West Islip, New York
  - Aesthetic Solutions /ID# 239074, Chapel Hill, North Carolina
  - Bellaire Dermatology Associates /ID# 239133, Bellaire, Texas

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible clinical trial data sharing. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: For details on when studies are available for sharing visit https://vivli.org/ourmember/abbvie/
Access Criteria: To learn more about the process, or to submit a request, visit the following link https://www.abbvieclinicaltrials.com/hcp/data-sharing/
URL: https://vivli.org/ourmember/abbvie/

REFERENCES:
- See also: Related Info — https://www.abbvieclinicaltrials.com/study/?id=2029-701-008